CLINICAL TRIAL: NCT03137537
Title: Ivabradine in the Management of Cardiac Autonomic Dysfunction Associated With Thoracic Radiation Therapy.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding terminated
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Anju Nohria, Assistant Professor in Internal Medicine, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-022
Record Dates: First submitted 2017-04-19; First posted 2017-05-02 (Actual); Results first posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Lymphoma; Autonomic Imbalance; Cancer Survivorship
Keywords: Lymphoma; Abnormal resting heart rate; Autonomic imbalance; Cancer survivorship
MeSH Terms: conditions — Lymphoma | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ivabradine (Experimental): * Ivabradine will be administered for a total of 6 weeks
  * Ivabradine is taken orally twice daily
  * Dosage will be adjusted according to physician determination
  Interventions: Drug: Ivabradine
- Placebo Oral Tablet (Placebo Comparator): * Placebo will be administered for a total of 6 weeks
  * Placebo is taken orally twice daily
  * Dosage will be adjusted according to physician determination
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Ivabradine — lower heart rate in heart failure patients.
  Other Names: Corlanor
  Arms: Ivabradine
Drug: Placebo Oral Tablet — Procedure prescribed to compare the active effect of a medicine.
  Arms: Placebo Oral Tablet

SUMMARY:
This study will explore whether ivabradine lowers heart rate, and thus improves exercise capacity, in survivors of lymphoma who have an elevated resting heart rate as a side effect of prior radiation treatment.

The drugs involved in this study are:

* Ivabradine
* Placebo

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

This research study is a Pilot Study, which is the first time investigators are examining this study intervention for this particular problem.

In this research study, the investigators are studying a drug called ivabradine. The investigators are exploring whether ivabradine can be used to reduce heart rate, increase exercise duration, and improve quality of life in survivors of lymphoma who received radiation to their chest as a part of their cancer treatment.

The U.S. Food and Drug Administration (FDA) has not approved ivabradine for this specific disease, but it has approved the drug as an oral medication to lower heart rate in heart failure patients.

Survivors of lymphoma who were treated with neck and/or chest radiation can have an elevated resting heart rate and an abnormal rate of decline in their heart rate after exercise, also known as cardiac autonomic dysfunction. These abnormalities can limit exercise duration and worsen quality of life in some radiation treated survivors of lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Survivors of mediastinal lymphoma (either Non-Hodgkin's Lymphoma or Hodgkin's Lymphoma) with no active malignancy
* Prior mediastinal or mantle radiation ≥ 5 years prior to enrollment in the study
* Age 18-80 years.
* Participants must have normal organ function as defined below:

  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine clearance ≥ 15 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* Normal sinus rhythm with resting heart rate ≥ 80 bpm on screening EKG
* Based on findings in animals, ivabradine may cause fetal harm when administered to a pregnant woman. For this reason, women of child-bearing potential must agree to use adequate contraception.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who are receiving any other investigational agents.
* History of allergic reaction to ivabradine.
* Participants receiving any medications or substances that are inhibitors or inducers of cytochrome P450 3A4 are ineligible.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, acute coronary syndrome, symptomatic known coronary artery disease, severe valvular heart disease, active malignancy, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because ivabradine is an agent with the potential for teratogenic effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ivabradine, breastfeeding should be discontinued if the mother is treated with ivabradine.
* HIV-positive participants on combination antiretroviral therapy.
* Patients with systolic blood pressure < 90 mm Hg.
* Patients with sick-sinus syndrome, sino-atrial block, third degree heart block, atrial fibrillation, and those with permanent pacemakers.
* Patients with other established indications for ivabradine: stable, symptomatic chronic HF with a left ventricular ejection fraction ≤ 35% and in sinus rhythm with a resting HR ≥ 70 bpm, who are taking maximally tolerated doses of beta-blockers or have contraindications to beta-blocker use.
* Patients with severe hepatic dysfunction (Child Pugh Class C).
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anju Nohria, MD, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ivabradine: * Ivabradine will be administered for a total of 6 weeks
  * Ivabradine is taken orally twice daily
  * Dosage will be adjusted according to physician determination
  Ivabradine: lower heart rate in heart failure patients.
- Placebo Oral Tablet: * Placebo will be administered for a total of 6 weeks
  * Placebo is taken orally twice daily
  * Dosage will be adjusted according to physician determination
  Placebo Oral Tablet: Procedure prescribed to compare the active effect of a medicine.
Period: Overall Study
Arm/Group | Ivabradine | Placebo Oral Tablet
Started | 12 | 11
Completed | 12 | 10
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivabradine | Placebo Oral Tablet | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Median (Full Range); unit: years] | 60 [45 to 70] | 52 [29 to 69] | 56 [29 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Beta-blocker at baseline [Count of Participants; unit: Participants] | 6 | 6 | 12
Ejection Fraction, % [Median (Full Range); unit: %] — Population: Baseline echo data not available in 2 pts randomized to the ivabradine group
  %
    number analyzed (Participants) | 10 | 11 | 21
    (all) | 61 [43 to 73] | 63 [50 to 69] | 63 [50 to 69]
Resting heart rate [Median (Full Range); unit: bpm] | 90 [76 to 104] | 93 [78 to 103] | 91 [76 to 104]

OUTCOME MEASURES:

1. Primary Outcome: To Investigate Whether Ivabradine Lowers Resting HR, Compared To Placebo, In Survivors Of Lymphoma
Description: Calculate the change in resting HR (from Holter monitor data) from baseline to 6 weeks for each patient in the study. Then compare the median change with ivabradine to the median change with placebo.
Time Frame: 6 weeks
Population: Analyzed all patients who had data available at baseline and at 6 weeks
Measure: Median (Full Range); unit: bpm
Arm/Group | Ivabradine | Placebo Oral Tablet
Number analyzed (Participants) | 12 | 10
bpm | -13 [-25 to 0] | -1 [-13 to 13]
Statistical Analysis 1: Comparison: Ivabradine vs Placebo Oral Tablet; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: To Evaluate Whether Ivabradine Improves Exercise Duration, Compared To Placebo, In Survivors Of Lymphoma
Description: Calculate the change in exercise duration (from exercise treadmill stress tests) from baseline to 6 weeks for each patient in the study. Then compare the median change in exercise duration with ivabradine to the median change in exercise duration with placebo.
Time Frame: 6 weeks
Measure: Median (Full Range); unit: minutes
Arm/Group | Ivabradine | Placebo Oral Tablet
Number analyzed (Participants) | 12 | 10
minutes | 0.4 [-2.7 to 2.6] | -0.1 [-1.0 to 0.9]
Statistical Analysis 1: Comparison: Ivabradine vs Placebo Oral Tablet; Test type: Superiority; p = 0.63, Wilcoxon (Mann-Whitney)

3. Other Pre Specified Outcome: To Evaluate Whether Ivabradine Improves Additional Markers of Cardiac Sympatho-vagal Balance, Compared To Placebo, In Survivors Of Lymphoma
Description: Calculate the change in cardiac autonomic function (from cardiac autonomic function testing) from baseline to 6 weeks in one half of the patients in the study (n=30)
Time Frame: 6 weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: To Evaluate Whether Ivabradine Improves Health Related Quality Of Life Compared To Placebo, In Survivors Of Lymphoma
Description: Calculate the change in health related quality of life (from SF-36 quality of life surveys) from baseline to 6 weeks for each patient in the study (n=60)
Time Frame: 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Ivabradine | Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 3/12 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivabradine (N=12) | Placebo Oral Tablet (N=11)
heart failure (Cardiac disorders) | 1 (1) | 0 (0)
sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 1 (1) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ankle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT03137537/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT03137537/ICF_001.pdf